CLINICAL TRIAL: NCT07286799
Title: Comparison of the Analgesic Efficacy of Posterior Quadratus Lumborum Block and Transversalis Fascia Plane Block in Children Undergoing Orchiopexy
Brief Title: Comparison of the Analgesic Efficacy of Transversalis Fascia Plane Block and Posterior Quadratus Lumborum Block in Pediatric Patient Undergoing Orchiopexy: A Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Reyhan Kucuk Erturk, Resident Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: E-48670771-514.9900
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Orchiopexy; Transversalis Fascia Plane Block; Quadratus Lumborum Block
Keywords: Transversalis fascia plane block; Quadratus lumborum block; Orchiopexy; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children aged 1-7 years undergoing orchiopexy who received a transversalis fascia plane block.: Children aged 1-7 years undergoing orchiopexy who received a transversalis fascia plane block.
- Children Aged 1-7 Years Undergoing Orchiopexy Who Received a Posterior Quadratus Lumborum Block: Children Aged 1-7 Years Undergoing Orchiopexy Who Received a Posterior Quadratus Lumborum Block

SUMMARY:
It was planned to compare the analgesic efficacy of the transversalis fascia plane block and the posterior quadratus lumborum block in children aged 1 to 7 years undergoing orchiopexy, by evaluating their FLACC scores and the time to first postoperative analgesic requirement.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 7 years with ASA physical status I-II undergoing unilateral orchiopexy surgery.

Exclusion Criteria:

* ASA physical status ≥ III
* History of prematurity (gestational age < 37 weeks) Known coagulation disorders or bleeding tendency
* Infection, inflammation, or skin lesion at the injection site
* Known neurological or neuromuscular diseases
* Presence of significant cardiac or pulmonary disease (e.g., congenital heart disease, active asthma)
* Hepatic or renal dysfunction
* Known allergy or hypersensitivity to local anesthetics (e.g., bupivacaine, lidocaine)
* Developmental delay or cognitive impairment that prevents accurate pain assessment
* Use of additional regional analgesia techniques (e.g., caudal block) during surgery
* Block failure or intraoperative complications requiring exclusion from protocol analysis
* Lack of parental consent for participation in the study

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1 to 7 years with ASA physical status I-II undergoing unilateral orchiopexy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Time to First Analgesic Requirement After Surgery | First 24 hours postoperatively
  The time elapsed from the end of surgery to the administration of the first rescue analgesic.

SECONDARY OUTCOMES:
FLACC Pain Scores at Specified Time Intervals | First 24 hours postoperatively
  Pain assessment using the Face, Legs, Activity, Cry, Consolability (FLACC) scale (score range: 0-10; higher scores indicate worse pain) at 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided